CLINICAL TRIAL: NCT04528381
Title: Role of Laparoscopy in Management of Non-palpable Undescended Testis : Assuit University Experience
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelfattah, Resident at genaral surgery department, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Laparoscopy in NPT
Record Dates: First submitted 2020-08-23; First posted 2020-08-27 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Undescended Testes
MeSH Terms: conditions — Cryptorchidism | interventions — Laparoscopy

STUDY DESIGN:
Intervention Model Description: Prospective & retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laparoscopy (Other): Diagnostic and therapeutic laparoscopy
  Interventions: Procedure: Laparoscopy

INTERVENTIONS:
Procedure: Laparoscopy — Laparoscopic orchiopexy

SUMMARY:
1. To evaluate the role of laparoscopy in diagnosis & treatment of Non- palpable undescended testis
2. To compare between different laparoscopic techniques
3. To introduce new laparoscopic technique in Assuit university " shehata technique "

DETAILED DESCRIPTION:
Cryptorchidism or undescended testis (UDT) is one of the most common genital anomalies in childhood. Its incidence is 3-5 % in full term newborn, and affect more than one third of premature newborn. The incidence decrease to 1 % at age of 3months. About 20% of UDT are impalpable, and about 50% of these impalpable testes are either vanished or atrophic (1-3).

Many diagnostic methods have been used for the evaluation and management of the undescended testis, including imaging studies and multiple surgical procedures.

Surgical management of UDT is performed to preserve testicular function (spermatogenesis) and to prevent the potential complications of undescended testis(1).

Regarding the optimal age of orchiopexy many recent findings suggest that early intervention (6 -12 months of age) is most beneficial. Other findings suggest that there is high rate of spontaneous descent during the first 3 months of life, so observation of undescended testis is advocated till 3 months of age, if the testis remains non-palpable at 3 months of age, it is unlikely to become palpable by waiting another 3 months. Therefore, diagnostic laparoscopy and orchidopexy could be performed from 3 months of age(2).

For intraabdominal cryptorchidism, laparoscopic surgery has been accepted by most surgeons as the preferred technique for diagnosis & treatment (4).

Laparoscopic findings in non-palpable testis include ; Absent testis either ; Agenesis ( absence of spermatic vessels and vas deferens ) or vanishing testis ( blind ending of spermatic vessels or vas ) , Canalicular testis ; Penetration of vas and spermatic vessels into the internal inguinal ring with or without directly seeing the testis , Abdominal testis Localized between the inferior renal pole and the ipsilateral internal inguinal ring. Can be low (< 2cm) or high (>2cm) from internal inguinal ring , Peeping ; Primarily in intra-abdominal position. The testis introduces itself into the inguinal canal due to the intra-abdominal pressure augmentation during the laparoscopic procedure.(5)

Several techniques have been described for treatment of intra-abdominal testis including microsurgical auto-transplantation, primary laparoscopic orchiopexy (VILO), one- and two-stage laparoscopic Fowler-Stephens procedures, and staged laparoscopic traction orchiopexy (Shehata technique

ELIGIBILITY:
Inclusion Criteria:

* any patient admitted to pediatric unit in Assuit University hospital with non palpable testis ( NPT )below age of 6 years

Exclusion Criteria:

* patients with NPT above age of 6 years
* patients with atrophic or vanishing testis
* patients with previous failed laparoscopic orchiopexy

Ages: 3 Months to 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Testicular volume | 3 months postoperative
  Achievement of near normal testicular volume
Testicular position | 3 months postoperative
  Achievement of of near normal testicular position (at scrotum )

SECONDARY OUTCOMES:
Postoperative complications | 3 months postoperative
  Bleeding , damage of vas and/or blood supply and reascent

REFERENCES:
- [Background] Elsherbeny M, Abdallah A, Abouzeid A, Ghanem W, Zaki A. Staged laparoscopic traction orchiopexy for intra-abdominal testis: Is it always feasible? J Pediatr Urol. 2018 Jun;14(3):267.e1-267.e4. doi: 10.1016/j.jpurol.2018.01.021. Epub 2018 Mar 2. PMID 29567012
- [Background] Shehata S, Shalaby R, Ismail M, Abouheba M, Elrouby A. Staged laparoscopic traction-orchiopexy for intraabdominal testis (Shehata technique): Stretching the limits for preservation of testicular vasculature. J Pediatr Surg. 2016 Feb;51(2):211-5. doi: 10.1016/j.jpedsurg.2015.10.063. Epub 2015 Nov 4. PMID 26655212
- [Background] Powell C, McIntosh J, Murphy JP, Gatti J. Laparoscopic orchiopexy for intra-abdominal testes-a single institution review. J Laparoendosc Adv Surg Tech A. 2013 May;23(5):481-3. doi: 10.1089/lap.2012.0578. Epub 2013 Apr 6. PMID 23560656